CLINICAL TRIAL: NCT06753305
Title: Evaluation of the Effect of Ozone Therapy Application on Wound Healing After Gingivoplasty
Brief Title: The Effect of Ozone Therapy on Gingivoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assoc. Prof. Dr., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-15/01
Record Dates: First submitted 2024-11-27; First posted 2024-12-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Gingival Enlargement
Keywords: Gingival enlargement; Ozone therapy; Wound healing; Gingivectomy; Gingivoplasty
MeSH Terms: conditions — Gingival Hyperplasia | interventions — Gingivectomy

STUDY DESIGN:
Intervention Model Description: The study will include 48 systemically healthy, systemically healthy patients older than 18 years of age, with gingival enlargement in the maxillary anterior region, requiring gingivectomy and gingivoplasty surgery, who applied to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology and İzmir Democracy University, Faculty of Dentistry, Department of Periodontology. Patients will be evaluated in two different groups as test and control group after surgery. Patients will be randomly allocated to the study groups by closed envelope method. The test group will receive periodontal paste (Coe-pak) + Ozone therapy (activated oxygen (Cure 09 Active Oxygen)) following gingivectomy and gingivoplasty surgery, while the control group will receive only periodontal paste application following gingivectomy and gingivoplasty surgery. All patients will undergo gingivectomy and gingivoplasty with the same procedure.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Other): Periodontal paste application (Coe-pak) using active oxygen (Cure 09 Active Oxygen) on the wound surface after gingivectomy and gingivoplasty surgery applied to the maxillary anterior regions
  Interventions: Procedure: Gingivectomy and gingivoplasty surgery and periodontal paste +ozone therapy application
- Control group (Other): Only periodontal paste application (Coe-pak) to the wound surface after gingivectomy and gingivoplasty surgery applied to the maxillary anterior regions
  Interventions: Procedure: Gingivectomy and gingivoplasty surgery and periodontal paste application

INTERVENTIONS:
Procedure: Gingivectomy and gingivoplasty surgery and periodontal paste +ozone therapy application — After taking systemic and dental anamnesis from all patients, Phase 1 periodontal treatment will be performed and oral hygiene education will be given. Patients will be called 4 weeks after treatment for re-evaluation and surgical treatment will be planned. After local anesthesia, the incision line will be determined with a marking press or periodontal probe according to the amount of gingival enlargement. An external bevel incision will be made along the determined incision line with a number 15 scalpel. After the incision is completed, the remaining tissues will be removed using microsurgical scissors. Then gingivoplasty will be performed. After gingivectomy and gingivoplasty, the surgical site will be left for secondary healing. Periodontal paste (Coe-pak) will be applied to the area left for secondary healing after ozone therapy (activated oxygen (Cure 09 Active Oxygen))
  Arms: Test group
Procedure: Gingivectomy and gingivoplasty surgery and periodontal paste application — After taking systemic and dental anamnesis from all patients, Phase 1 periodontal treatment will be performed and oral hygiene education will be given. Patients will be called 4 weeks after treatment for re-evaluation and surgical treatment will be planned. After local anesthesia, the incision line will be determined with a marking press or periodontal probe according to the amount of gingival enlargement. An external bevel incision will be made along the determined incision line with a number 15 scalpel. After the incision is completed, the remaining tissues will be removed using microsurgical scissors. Then gingivoplasty will be performed. After gingivectomy and gingivoplasty, the surgical site will be left for secondary healing. Only periodontal paste will be applied after the surgery.
  Arms: Control group

SUMMARY:
Ozone therapy after gingivectomy and gingivoplasty has been found to reduce patients' pain levels and positively impact their quality of life. This study aimed to compare the healing potential of the wound surface following gingivectomy and gingivoplasty surgery applied to the maxillary anterior regions with classical periodontal paste application (Coe-pak) using activated oxygen (Cure 09 Active Oxygen) and classical periodontal paste application only (Coe-pak).

The study will include 48 systemically healthy patients older than 18 years of age with gingival enlargement in the maxillary anterior region, requiring gingivectomy and gingivoplasty surgery, who applied to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology and Izmir Democracy University, Faculty of Dentistry, Department of Periodontology. Patients will be evaluated in two different groups as test and control group after surgery. Patients will be randomly divided into study groups by closed envelope method. The test group will receive periodontal paste (Coe-pak) + Ozone therapy (active oxygen (Cure 09 Active Oxygen)) after gingivectomy and gingivoplasty surgery, while the control group will receive only periodontal paste after gingivectomy and gingivoplasty surgery. All patients will undergo gingivectomy and gingivoplasty with the same procedure

DETAILED DESCRIPTION:
Gingival enlargement leads to unaesthetic appearance, increased susceptibility to periodontal disease and halitosis by making it difficult to control plaque, and chewing and speech disorders by affecting functional function. Gingivectomy and gingivoplasty are used for the excision of diseased gingiva or gingival enlargement to create a natural anatomical form of the gingiva and improve aesthetics. After gingivectomy and gingivoplasty surgery, secondary healing occurs at the wound site. Bleeding and pain as a result of secondary healing negatively affect the patient's quality of life. Many different treatment methods such as ozone therapy, laser therapy, antiseptic agents, platelet concentrate, and herbal products are applied to reduce postoperative complications and increase patient comfort after gingivectomy and gingivoplasty. Since ozone gas increases growth factors, activates local antioxidant mechanisms, and supports tissue repair, its application to the wound site prevents postoperative infection and may accelerate wound healing. Topical application of ozone gas has been reported to be effective in the early stages of wound healing by increasing the amount of vascular endothelial growth factor expression. In a systematic review aiming to evaluate the effectiveness of ozone therapy in reducing the symptoms of oral diseases, especially oral mucositis, which is a serious complication of cancer treatment, it was confirmed that ozone has analgesic, anti-inflammatory, antimicrobial, and regenerative properties. In a study, it was found that the application of ozone therapy after gingivectomy and gingivoplasty reduced the pain levels of patients and positively affected their quality of life. To compare the healing potential of the wound surface following gingivectomy and gingivoplasty surgery applied to the maxillary anterior regions with the application of classical periodontal paste (Coe-pak) using activated oxygen (Cure 09 Active Oxygen) and with the application of classical periodontal paste (Coe-pak) alone.

The study will include 48 systemically healthy, systemically healthy patients older than 18 years of age, with gingival enlargement in the maxillary anterior region, requiring gingivectomy and gingivoplasty surgery, who applied to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology and İzmir Democracy University, Faculty of Dentistry, Department of Periodontology. All patients will be called for re-evaluation 4 weeks after phase 1 periodontal treatment and surgical treatment will be planned. Clinical measurements (plaque index, gingival index, pocket depth, bleeding index on probing, and gingival overgrowth index) and oral health impact profile-14 questionnaire will be recorded and standard photographs will be taken before surgery. After local anesthesia, the incision line will be determined with a marking press or periodontal probe according to the amount of gingival enlargement. An external beveled incision will be made along the determined incision line with a No. 15 scalpel. Once the incision is complete, the surrounding tissues will be cleaned using microsurgical scissors. Following this, gingivoplasty will be performed. Patients will be randomly assigned to either the test group or the control group. In the test group, periodontal paste (Coe-Pak) will be applied to the area designated for secondary healing after ozone therapy (Cure 09 Active Oxygen). In the control group, only periodontal paste (Coe-Pak) will be applied. Postoperatively, the patient will record the bleeding status, daily analgesic use, and pain and burning with a visual analog scale for the first 7 days. Standard photographs will be taken in the postoperative period, immediately after the placement of the patch and on the 7th, 14th and 21st days. In addition, clinical evaluations (healing index, inflammation, modified manchester scar scale, surgical Area Plaque index, re-epithelialisation evaluation, and only on the 7th day, plaque accumulation in the periodontal paste) will be recorded from the patients on the 7th, 14th, and 21st days.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years old
2. Systemically healthy individuals
3. Gingival enlargement due to inflammation in at least 4 teeth in the maxillary anterior region
4. Horizontal and vertical gingival growth index score of 1 or 2
5. Gingival thickness more than 2 mm
6. Good oral hygiene
7. No loss of clinical attachment

Exclusion Criteria:

1. Pregnancy
2. Hereditary gingival fibromatosis
3. Drug-induced gingival enlargement
4. Allergy
5. Presence of systemic conditions requiring antibiotic prophylaxis
6. Acute and untreated periodontitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Gingival inflammation | 1-month follow-up after gingivectomy and gingivoplasty surgery
  The effect of ozone therapy on inflammation will be measured in the 1-month follow-up after gingivectomy and gingivoplasty surgery.
  Inflammation 0=no inflammation,
  1. mild inflammation,
  2. moderate inflammation,
  3. severe inflammation
Gingival contour | 1-month follow-up after gingivectomy and gingiplasty
  The effect of ozone therapy on gingival contour after gingivectomy and gingivoplasty surgery was measured using the Modified Manchester Scar Scale at 1-month follow-up.
  Modified Manchester Scar Scale (used to assess gingival colour, contour, and distortion) The colour of the wound compared to the adjacent mucosa score 0= perfect fit score 1= slight non-compliance score 2= obvious incompatibility The contour of the wound compared to the surrounding tissues score 0= similar score 1= slightly raised or indented score 2= hypertrophic Wound distortion score 0= no distortion score 1= slight distortion score 2= obvious distortion The total of the scores in the three categories indicates the wound healing score, the total score ranges from 0 to 6, with lower scores indicating better healing.
Re-epithelialisation evaluation | 1-month follow-up after gingivectomy and gingivoplasty surgery
  To measure the effect of ozone therapy on re-epithelialization after gingivectomy and gingivoplasty surgeries with toluidine blue or 3% H2O2 intraoral photographs at 1-month follow-up.
Gingival distortion | 1-month follow-up after gingivectomy and gingiplasty
  To measure the effect of ozone therapy on gingival distorrion via Modified Manchester Scar Scale after gingivectomy and gingivoplasty surgery at 1-month follow-up.
  Modified Manchester Scar Scale (used to assess gingival colour, contour, and distortion) The colour of the wound compared to the adjacent mucosa score 0= perfect fit score 1= slight non-compliance score 2= obvious incompatibility The contour of the wound compared to the surrounding tissues score 0= similar score 1= slightly raised or indented score 2= hypertrophic Wound distortion score 0= no distortion score 1= slight distortion score 2= obvious distortion The total of the scores in the three categories indicates the wound healing score, the total score ranges from 0 to 6, with lower scores indicating better healing.

SECONDARY OUTCOMES:
Patient's quality of life | 1-month follow-up after gingivectomy and gingiplasty
  The effect of ozone therapy on wound healing after gingivectomy and gingivoplasty surgery will be measured at 1-month follow-up using a visual analog scale on patient quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler Ayyıldız, Assoc. Prof., Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
  Statistical Analysis Plan (SAP)
Supporting Information: Study Protocol, SAP
Time Frame: The work will be shared 6 months after publication
Access Criteria: It will be shared in case the principal investigator is contacted.

REFERENCES:
- [Background] Uslu MO, Akgul S. Evaluation of the effects of photobiomodulation therapy and ozone applications after gingivectomy and gingivoplasty on postoperative pain and patients' oral health-related quality of life. Lasers Med Sci. 2020 Sep;35(7):1637-1647. doi: 10.1007/s10103-020-03037-8. Epub 2020 May 20. PMID 32435906
- [Background] Gupta G, Mansi B. Ozone therapy in periodontics. J Med Life. 2012 Feb 22;5(1):59-67. Epub 2012 Mar 5. PMID 22574088
- [Background] Eroglu ZT, Kurtis B, Altug HA, Sahin S, Tuter G, Baris E. Effect of topical ozonetherapy on gingival wound healing in pigs: histological and immuno-histochemical analysis. J Appl Oral Sci. 2018 Dec 10;27:e20180015. doi: 10.1590/1678-7757-2018-0015. PMID 30540068
- [Background] Chesterman J, Beaumont J, Kellett M, Durey K. Gingival overgrowth: Part 2: management strategies. Br Dent J. 2017 Feb 10;222(3):159-165. doi: 10.1038/sj.bdj.2017.111. PMID 28184072
- [Background] Bozkurt E, Uslu MO. Evaluation of the effects of platelet-rich fibrin, concentrated growth factors, and autologous fibrin glue application on wound healing following gingivectomy and gingivoplasty operations: a randomized controlled clinical trial. Quintessence Int. 2022 Mar 14;53(4):328-341. doi: 10.3290/j.qi.b2449819. PMID 34927405
- [Background] Kusakci-Seker B, Demirayak-Akdemir M. The effect of non-thermal atmospheric pressure plasma application on wound healing after gingivectomy. Int Wound J. 2020 Oct;17(5):1376-1383. doi: 10.1111/iwj.13379. Epub 2020 May 27. PMID 32462820
- [Background] Beaumont J, Chesterman J, Kellett M, Durey K. Gingival overgrowth: Part 1: aetiology and clinical diagnosis. Br Dent J. 2017 Jan 27;222(2):85-91. doi: 10.1038/sj.bdj.2017.71. PMID 28127024